CLINICAL TRIAL: NCT01123590
Title: Characteristics of Patients With Thymoma Undergone Thymectomy in Chulalongkorn Hospital Between 2003-2007
Brief Title: Characteristics of Patients With Thymoma in Chulalongkorn Hospital
Status: Completed | Type: Observational
Sponsor: Chulalongkorn University (Other)
Responsible Party: Jettanong Klaewsongkram, Chulalongkorn University
Other Study IDs: Chula-ARC 003/09
Record Dates: First submitted 2010-05-12; First posted 2010-05-14 (Estimated); Last update posted 2010-11-23 (Estimated); Status verified 2010-11

CONDITIONS: Thymoma Staging; Clinical Presentations; Associated Disorders; Laboratory Findings
Keywords: Thymoma; Autoimmune diseases; Immunodeficiency
MeSH Terms: conditions — Thymoma; Autoimmune Diseases; Immunologic Deficiency Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — PBMC
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Thymoma: Patients with thymoma
- Control: Normal controls

SUMMARY:
The purpose of this study is to study characteristics of patients with thymoma in Chulalongkorn hospital between 2003-2007.

DETAILED DESCRIPTION:
To study characteristics of patients with thymoma undergone thymectomy in Chulalongkorn hospital between 2003-2007 in terms of clinical manifestations, associated diseases, and laboratory findings.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histocytological proved thymoma undergone thymectomy in Chulalongkorn hospital between 2003-2007

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with thymoma undergone thymectomy in Chulalongkorn hospital between 2003-2007
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2009-11; Primary Completion 2010-04 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Thymoma staging and clinical manifestations | 5 years

SECONDARY OUTCOMES:
Associated diseases and laboratory findings Immunological data | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Jettanong Klaewsongkram, MD, Principal Investigator — Chulalongkorn University
Locations (1):
- Faculty of Medicine, Chulalongkorn University, Bangkok, Thailand

REFERENCES:
- [Derived] Thongprayoon C, Tantrachoti P, Phatharacharukul P, Buranapraditkun S, Klaewsongkram J. Associated immunological disorders and cellular immune dysfunction in thymoma: a study of 87 cases from Thailand. Arch Immunol Ther Exp (Warsz). 2013 Feb;61(1):85-93. doi: 10.1007/s00005-012-0207-9. Epub 2012 Dec 11. PMID 23229679